CLINICAL TRIAL: NCT01931722
Title: Can Branched Chained Amino Acid Supplementation Combined With Strength-Training Minimize Sarcopenia in Older Men?
Brief Title: Exercise and Branched Chain Amino Acids (BCAA)Requirements in Older Men
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: not able to find enough participants for this study
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Professor and Weider Research Chair, University of Western Ontario, Canada
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 002
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Sarcopenia
Keywords: branched chain amino acid requirement; older men; strength training; sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Amino Acids, Branched-Chain; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Branched chain amino acid (Active Comparator): Branched chain amino acid as food supplement
  Interventions: Dietary Supplement: Branched chain amino acid; Behavioral: Strength training
- Weight training (Active Comparator): Strength training will include a split-training program using all major muscle groups of the body on a three day "on", one day "off" protocol. Muscle areas targeted on each training day will be as follows: Day1: chest, shoulder, triceps; Day2: back, biceps; Day3: legs and calfs; Day4: will be a rest day. On Day5: this cycle will begin again. A combination of free weights and machines will be used for each training day. Progressive overload protocol will be applied where the load used by every participant will be adjusted bi-weekly based on their 70% of 1RM (repetition maximum). Instruction will be provided for all exercises and professional trainers will oversee all training sessions.
  Interventions: Dietary Supplement: Branched chain amino acid; Behavioral: Strength training

INTERVENTIONS:
Dietary Supplement: Branched chain amino acid — seven graded intakes of a BCAA (branched chain amino acid) mixture from 50 to 350 mg.kg-1.d-1 will be used to measure BCAA requirement
  Other Names: Ajinomoto branched chain amino acids
Behavioral: Strength training — Strength training will include a split-training program using all major muscle groups of the body on a three day "on", one day "off" protocol. Muscle areas targeted on each training day will be as follows: Day1: chest, shoulder, triceps; Day2: back, biceps; Day3: legs and calfs; Day4: will be a rest day. On Day5: this cycle will begin again. A combination of free weights and machines will be used for each training day. Progressive overload protocol will be applied where the load used by every participant will be adjusted bi-weekly based on their 70% of 1 repetition maximum (maximum weight that can be lifted only one time). Instruction will be provided for all exercises and professional trainers will oversee all training sessions.
  Other Names: weight training

SUMMARY:
Likely, branched chain amino acid (BCAA) requirements are increased in older strength-trained (ST) individuals. If so, supplementation in this group will maximize muscle protein synthesis (MPS) and minimize loss of muscle with age (sarcopenia).

DETAILED DESCRIPTION:
We hypothesize that the dietary requirement for the branched chain amino acids (BCAA) in an older strength-trained (ST) population will be greater than the current recommendation (RDA). If so, a greater intake of BCAA together with ST is necessary if one aims to maximize muscle protein synthesis (MPS). Currently, the BCAA requirement in the ST older population (55-65 y) is unknown. This is critical information especially given the value of ST for overall health.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active (~2-3 h/wk of physical activity) healthy older men (55-65 y)
* A minimum of 4 month weight training experience

Exclusion Criteria:

* Have symptoms or take medication for respiratory disease
* Have symptoms or take medication for cardiovascular disease
* Have symptoms or take medication for metabolic disease
* Have symptoms or take mediation for neuromuscular disease
* Use heart rate or blood pressure medications
* Use any medications with side effects of dizziness, lack of motor control, or slowed reaction time
* Have an excessive alcohol intake (more than 2 drinks per day)
* Have any cardiovascular or neuromuscular limitations to exercise
* Are allergic to milk or milk products
* Use anabolic steroids or performance enhancing drugs

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Required Branched chain amino acid of older strength trained men | 12 months
  Branched chain amino acid requirement will be measured in 55-65 years old strength trained men using indicator amino acid oxidation method

SECONDARY OUTCOMES:
Muscle size | 12 months
  cross-sectional measure of muscle size will be measured in all participants using standard procedures of magenetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — The University of Western Ontario; Arash Bandegan, MSc., Study Director — The University of Western Ontario
Locations (1):
- Exercise Nutrition Research Laboratory, London, Ontario, Canada

REFERENCES:
- [Background] Riazi R, Wykes LJ, Ball RO, Pencharz PB. The total branched-chain amino acid requirement in young healthy adult men determined by indicator amino acid oxidation by use of L-[1-13C]phenylalanine. J Nutr. 2003 May;133(5):1383-9. doi: 10.1093/jn/133.5.1383. PMID 12730426
- [Background] Lemon PW, Tarnopolsky MA, MacDougall JD, Atkinson SA. Protein requirements and muscle mass/strength changes during intensive training in novice bodybuilders. J Appl Physiol (1985). 1992 Aug;73(2):767-75. doi: 10.1152/jappl.1992.73.2.767. PMID 1400008
- [Background] Norton LE, Layman DK. Leucine regulates translation initiation of protein synthesis in skeletal muscle after exercise. J Nutr. 2006 Feb;136(2):533S-537S. doi: 10.1093/jn/136.2.533S. PMID 16424142
- [Background] Pencharz PB, Ball RO. Different approaches to define individual amino acid requirements. Annu Rev Nutr. 2003;23:101-16. doi: 10.1146/annurev.nutr.23.011702.073247. Epub 2003 Feb 21. PMID 12626690
- [Background] Volpi E, Kobayashi H, Sheffield-Moore M, Mittendorfer B, Wolfe RR. Essential amino acids are primarily responsible for the amino acid stimulation of muscle protein anabolism in healthy elderly adults. Am J Clin Nutr. 2003 Aug;78(2):250-8. doi: 10.1093/ajcn/78.2.250. PMID 12885705
- [Background] Lemon PW. Beyond the zone: protein needs of active individuals. J Am Coll Nutr. 2000 Oct;19(5 Suppl):513S-521S. doi: 10.1080/07315724.2000.10718974. PMID 11023001
- [Background] Layman DK, Walker DA. Potential importance of leucine in treatment of obesity and the metabolic syndrome. J Nutr. 2006 Jan;136(1 Suppl):319S-23S. doi: 10.1093/jn/136.1.319S. PMID 16365106
- [Background] Kim JS, Wilson JM, Lee SR. Dietary implications on mechanisms of sarcopenia: roles of protein, amino acids and antioxidants. J Nutr Biochem. 2010 Jan;21(1):1-13. doi: 10.1016/j.jnutbio.2009.06.014. Epub 2009 Oct 1. PMID 19800212
- [Background] Katsanos CS, Kobayashi H, Sheffield-Moore M, Aarsland A, Wolfe RR. A high proportion of leucine is required for optimal stimulation of the rate of muscle protein synthesis by essential amino acids in the elderly. Am J Physiol Endocrinol Metab. 2006 Aug;291(2):E381-7. doi: 10.1152/ajpendo.00488.2005. Epub 2006 Feb 28. PMID 16507602
- [Background] Katsanos CS, Kobayashi H, Sheffield-Moore M, Aarsland A, Wolfe RR. Aging is associated with diminished accretion of muscle proteins after the ingestion of a small bolus of essential amino acids. Am J Clin Nutr. 2005 Nov;82(5):1065-73. doi: 10.1093/ajcn/82.5.1065. PMID 16280440
- [Background] Humayun MA, Elango R, Ball RO, Pencharz PB. Reevaluation of the protein requirement in young men with the indicator amino acid oxidation technique. Am J Clin Nutr. 2007 Oct;86(4):995-1002. doi: 10.1093/ajcn/86.4.995. PMID 17921376
- [Background] Dardevet D, Rieu I, Fafournoux P, Sornet C, Combaret L, Bruhat A, Mordier S, Mosoni L, Grizard J. Leucine: a key amino acid in ageing-associated sarcopenia? Nutr Res Rev. 2003 Jun;16(1):61-70. doi: 10.1079/NRR200252. PMID 19079937
- [Background] Cermak NM, Res PT, de Groot LC, Saris WH, van Loon LJ. Protein supplementation augments the adaptive response of skeletal muscle to resistance-type exercise training: a meta-analysis. Am J Clin Nutr. 2012 Dec;96(6):1454-64. doi: 10.3945/ajcn.112.037556. Epub 2012 Nov 7. PMID 23134885
- [Background] Bross R, Ball RO, Pencharz PB. Development of a minimally invasive protocol for the determination of phenylalanine and lysine kinetics in humans during the fed state. J Nutr. 1998 Nov;128(11):1913-9. doi: 10.1093/jn/128.11.1913. PMID 9808642
- [Background] Campbell WW, Trappe TA, Wolfe RR, Evans WJ. The recommended dietary allowance for protein may not be adequate for older people to maintain skeletal muscle. J Gerontol A Biol Sci Med Sci. 2001 Jun;56(6):M373-80. doi: 10.1093/gerona/56.6.m373. PMID 11382798